CLINICAL TRIAL: NCT06167304
Title: Digital Home Exercise Program Versus Standard of Care for Chronic OA-related Knee Pain: a Non-inferiority Randomized Controlled Trial
Brief Title: Physical Therapy vs Remote Exercise for Knee Pain Due to Osteoarthritis (OA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor halted funding
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-22-01430
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis; Chronic Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Technology-implemented exercise therapy (Experimental): Therapy plans performed at home overseen by a remote physical therapist via SimpleTherapy. Allocation to this group will require using smart devices or a computer/laptop to receive care. Remote visits with a PT typically last 45min long and home exercises suggested by the app are self-paced.
  Interventions: Other: Technology-implemented exercise therapy
- Traditional Physical Therapy (Active Comparator): Participants will be prescribed an exercise plan by a physical therapist as normally would occur as part of standards of care outside the context of a research study. In-person assessments and at-home exercise suggestions will be decided by the physical therapist. Duration of PT appointments is typically 45 minutes long two times per week and are supplemented by PT recommended self-paced at-home exercises.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Other: Technology-implemented exercise therapy — Therapy plans are performed at home overseen by a remote physical therapist via SimpleTherapy.
  Arms: Technology-implemented exercise therapy
Other: Traditional Physical Therapy — Traditional physical therapy per Standard of care.
  Arms: Traditional Physical Therapy

SUMMARY:
The purpose of this clinical study is to demonstrate that after six weeks of at home exercise, 3 times per week with SimpleTherapy, participants with clinical indications of knee OA will on average have improved outcomes noninferior than traditionally prescribed physical therapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Living in the tristate area - CT/NY/NJ
* Symptomatic OA (National Institute for Health and Care Excellence clinical criteria for OA)
* Chronic knee pain (>3 months) as a primary pain complaint
* Average pain score ≥ 4 on an 11-point numeric rating scale at baseline
* Access to a device with internet connection
* KL Stages 1-2-3

Exclusion Criteria:

* Prior documented history of cognitive impairment;
* History of total knee arthroplasty;
* History of: Inflammatory arthritis (e.g. rheumatoid arthritis); or any neuropathies affecting the lower limbs, spinal cord injury, spine fractures, advanced heart disease, bleeding issues (i.e. hemophilia), surgery within the last 90 days; fall within 90 days; high risk of fracture;
* History of knee injury, within the last 3 months;
* Currently engaged with other PT or strengthening program;
* Present unstable/uncontrolled cardiovascular condition
* Undergoing active chemotherapy for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline Week 0
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales rated 0-4, with higher score indicating more severe knee problems: symptoms, pain, activities of daily living (ADLs), sports/recreation, and quality of life. Full scale from 0-100, with higher score indicating more severe knee problems.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline Week 2
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales rated 0-4, with higher score indicating more severe knee problems: symptoms, pain, ADLs, sports/recreation, and quality of life. Full scale from 0-100, with higher score indicating more severe knee problems.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales rated 0-4, with higher score indicating more severe knee problems: symptoms, pain, ADLs, sports/recreation, and quality of life. Full scale from 0-100, with higher score indicating more severe knee problems.

SECONDARY OUTCOMES:
Brief Pain Inventory - short form (BPI-SF) | Baseline Week 0
  The BPI -SF rates severity pain and the degree to which pain interferes with common dimensions of feeling and function. It includes 9 items (0-No pain to 10-Pain as bad as you can imagine) and results in two scores ranging between 0-10: Pain Intensity and Pain Interference, with higher score indicating worse outcomes.
Brief Pain Inventory | Baseline Week 2
  The BPI -SF rates severity pain and the degree to which pain interferes with common dimensions of feeling and function. It includes 9 items (0-No pain to 10-Pain as bad as you can imagine) and results in two scores ranging between 0-10: Pain Intensity and Pain Interference, with higher score indicating worse outcomes.
Brief Pain Inventory | 12 weeks
  The BPI -SF rates severity pain and the degree to which pain interferes with common dimensions of feeling and function. It includes 9 items (0-No pain to 10-Pain as bad as you can imagine) and results in two scores ranging between 0-10: Pain Intensity and Pain Interference, with higher score indicating worse outcomes.
Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline Week 0
  Measures are based on "item banks," sets of items that represent symptom or functional domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. The T-score is provided with an error term (Standard Error or SE, 95% confidence interval).
Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline Week 2
  Measures are based on "item banks," sets of items that represent symptom or functional domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. The T-score is provided with an error term (Standard Error or SE, 95% confidence interval).
Patient Reported Outcomes Measurement Information System (PROMIS) | 12 weeks
  Measures are based on "item banks," sets of items that represent symptom or functional domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. The T-score is provided with an error term (Standard Error or SE, 95% confidence interval).
PSEQ-2 (Pain Self efficacy questionnaire-SF 2) | Baseline Week 0
  Assesses pain self-efficacy, which is a belief in one's ability to carry out activities even when in pain. The PSEQ-2 is a shorter version of PROMISE Self-Efficacy for Managing Chronic pain and it has been clinically validated. PSEQ-2 includes two items scored on a 7-point Likert scale (0- not at all confident to 6- Completely confident) which are added to form a total score ranging from 0 to 12. High scores indicate greater self-efficacy.
PSEQ-2 (Pain Self efficacy questionnaire-SF 2) | Baseline Week 2
  Assesses pain self-efficacy, which is a belief in one's ability to carry out activities even when in pain. The PSEQ-2 is a shorter version of PROMISE Self-Efficacy for Managing Chronic pain and it has been clinically validated. PSEQ-2 includes two items scored on a 7-point Likert scale (0- not at all confident to 6- Completely confident) which are added to form a total score ranging from 0 to 12. High scores indicate greater self-efficacy.
PSEQ-2 (Pain Self efficacy questionnaire-SF 2) | 12 weeks
  Assesses pain self-efficacy, which is a belief in one's ability to carry out activities even when in pain. The PSEQ-2 is a shorter version of PROMISE Self-Efficacy for Managing Chronic pain and it has been clinically validated. PSEQ-2 includes two items scored on a 7-point Likert scale (0- not at all confident to 6- Completely confident) which are added to form a total score ranging from 0 to 12. High scores indicate greater self-efficacy.
Work Productivity and Activity Impairment (WPAI) | Baseline Week 0
  WPAI measures impairments in work and activities. The WPAI yields four types of scores:
  A. Absenteeism B. Presenteeism C. Work productivity loss (overall work impairment / absenteeism plus presenteeism; D. Activity Impairment
  WPAI outcomes are expressed as impairment percentages (0%-100%), with higher numbers indicating greater impairment and less productivity (worse outcomes).
Work Productivity and Activity Impairment (WPAI) | Baseline Week 2
  WPAI measures impairments in work and activities. The WPAI yields four types of scores:
  A. Absenteeism B. Presenteeism C. Work productivity loss (overall work impairment / absenteeism plus presenteeism; D. Activity Impairment
  WPAI outcomes are expressed as impairment percentages (0%-100%), with higher numbers indicating greater impairment and less productivity (worse outcomes).
Work Productivity and Activity Impairment (WPAI) | 12 weeks
  WPAI measures impairments in work and activities. The WPAI yields four types of scores:
  A. Absenteeism B. Presenteeism C. Work productivity loss (overall work impairment / absenteeism plus presenteeism; D. Activity Impairment
  WPAI outcomes are expressed as impairment percentages (0%-100%), with higher numbers indicating greater impairment and less productivity (worse outcomes).
PGI-C (Patient global impression of change) | Baseline Week 0
  Captures perception of change in activity, limitations, feelings, emotions and health related QOL related to pain. PGIC is a 7 point scale depicting a patient's overall improvement rating. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." Measure correlations of patient ratings of importance of change with the magnitude of that change. The PGI-I is a transition scale that is a single question asking the patient to rate their condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.
PGI-C (Patient global impression of change) | Baseline Week 2
  Captures perception of change in activity, limitations, feelings, emotions and health related QOL related to pain. PGIC is a 7 point scale depicting a patient's overall improvement rating. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." Measure correlations of patient ratings of importance of change with the magnitude of that change. The PGI-I is a transition scale that is a single question asking the patient to rate their condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.
PGI-C (Patient global impression of change) | 12 weeks
  Captures perception of change in activity, limitations, feelings, emotions and health related QOL related to pain. PGIC is a 7 point scale depicting a patient's overall improvement rating. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." Measure correlations of patient ratings of importance of change with the magnitude of that change. The PGI-I is a transition scale that is a single question asking the patient to rate their condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.
Tampa Kinesiophobia Scale (TSK) | Baseline Week 0
  TSK is a self-reported questionnaire that quantifies fear of movement, or (re)injury. Individual item scores range from 1-4, with the negatively worded items having a reverse scoring. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Tampa Kinesiophobia Scale | Baseline Week 2
  TSK is a self-reported questionnaire that quantifies fear of movement, or (re)injury. Individual item scores range from 1-4, with the negatively worded items having a reverse scoring. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Tampa Kinesiophobia Scale | 12 weeks
  TSK is a self-reported questionnaire that quantifies fear of movement, or (re)injury. Individual item scores range from 1-4, with the negatively worded items having a reverse scoring. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Pain Catastrophizing Scale | Baseline Week 0
  13-item self reported measure designed to assess catastrophic thinking related to pain among adults. Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Pain Catastrophizing Scale | Baseline Week 2
  13-item self reported measure designed to assess catastrophic thinking related to pain among adults. Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Pain Catastrophizing Scale | 12 weeks
  13-item self reported measure designed to assess catastrophic thinking related to pain among adults. Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Subjective questionnaire (ST arm) | 12 weeks
  6-item questionnaire (yes/no) assessing accessibility, satisfaction with care and pain management, enjoyment, referral to friends or colleagues, and one open answer on recommendations for the exercise intervention.
Medication (PT arm) | 12 weeks
  Questionnaire asking Yes/No for starting new prescribed medication or treatment (if yes, name of new medication/treatment is requested).
Difficulty of exercises (PT arm) | 12 weeks
  Questionnaire tracking difficulty of exercises (0-not difficult at all, to 10- Extremely Difficult), total score ranges 0-10, with higher scores indicating greater difficulty.
Number of exercises completed (PT arm) | 12 weeks
  Questionnaire tracking home exercise adherence (How many Exercises this week?).

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Abilities Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only sharing analyzed deidentified information, not individual participant data.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT06167304/ICF_000.pdf